CLINICAL TRIAL: NCT06724120
Title: Construction of an Artificial Intelligence Prognostic Prediction Model for Sepsis Based on Time Series Analysis
Brief Title: Artificial Intelligence Prognostic Model for Sepsis Based on Time Series Analysis
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chi Zhang, Dr. Chi Zhang, West China Hospital
Other Study IDs: No.126 in 2024
Record Dates: First submitted 2024-11-30; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Sepsis; Prognostic Model; Artificial Intelligence; Individuality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survival Group
  Interventions: Other: No interventions
- Non-survival Group
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. It is one of the leading causes of death and disability worldwide, with an inpatient mortality rate of 10-20%. Sepsis is a severe complication in critically ill patients and can lead to septic shock and multiple organ dysfunction syndrome (MODS), usually triggered by severe trauma, surgery, and infections. Despite the availability of advanced diagnostic, therapeutic, and monitoring technologies, the incidence and mortality of sepsis remain high, posing a significant global challenge to the medical community. Over 49 million people worldwide develop sepsis annually, with approximately 11 million deaths, resulting in a mortality rate of about 15%-25%.

This study aims to develop a prognosis prediction model for sepsis patients using a neural network architecture (Transformer algorithm), based on time-series data. The primary outcome observed is the mortality outcome of sepsis patients. The goal of the research is to enhance the early identification of high-risk sepsis patients, thereby optimizing the timing of sepsis treatment and intervention and improving the accuracy of prognosis prediction for sepsis patients.

DETAILED DESCRIPTION:
1. Research Background Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. It is one of the leading causes of death and disability worldwide, with an inpatient mortality rate of 10-20%. Sepsis is a severe complication in critically ill patients and can lead to septic shock and multiple organ dysfunction syndrome (MODS), usually triggered by severe trauma, surgery, and infections. Despite the availability of advanced diagnostic, therapeutic, and monitoring technologies, the incidence and mortality of sepsis remain high, posing a significant global challenge to the medical community. Over 49 million people worldwide develop sepsis annually, with approximately 11 million deaths, resulting in a mortality rate of about 15%-25%.

2. Research Objectives and Content

1. Research Objective This study aims to develop a prognosis prediction model for sepsis patients using a neural network architecture (Transformer algorithm), based on time-series data. The primary outcome observed is the mortality outcome of sepsis patients. The goal of the research is to enhance the early identification of high-risk sepsis patients, thereby optimizing the timing of sepsis treatment and intervention and improving the accuracy of prognosis prediction for sepsis patients.
2. Research Content 2.1 Inclusion Criteria Patients diagnosed with sepsis at West China Hospital of Sichuan University from January 2020 to December 2023.

   2.2 Exclusion Criteria 1) Age under 18 years; 2) Gender unknown; 3) Incorrect or invalid discharge diagnosis; 4) Hospitalization period less than 24 hours; 5) Missing data exceeds 30%. 2.3 Sample Size 3,000 cases. 2.4 Data to be Collected A retrospective analysis of the clinical data of patients diagnosed with sepsis at West China Hospital of Sichuan University from January 2020 to December 2023 will be conducted. The baseline data of patients (including age, gender, comorbidities, history of malignant tumors, lesion sites, pathological types, etc.), occurrence of severe complications, total hospital stay, survival time, and other relevant information will be summarized to build a time-series-based prognosis prediction model for sepsis mortality risk.
3. Clinical Research Ethical Principles and Requirements This clinical research will comply with the Declaration of Helsinki issued by the World Medical Association and the relevant regulations set forth by the National Health and Family Planning Commission of the People's Republic of China concerning the Ethical Review of Biomedical Research Involving Human Subjects. The research will only utilize retrospective medical records and/or specimens, with all personal identifiers removed. There will be no risk to the subjects, nor will it negatively impact their rights or health. Therefore, informed consent is waived. The research data will be stored at West China Hospital of Sichuan University, accessible to the researchers, supervising departments, and the ethics review committee. Any public reports related to the research findings will not disclose the personal identity of the subjects. We will make every effort within the legal framework to protect the privacy and personal medical information of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with sepsis at West China Hospital of Sichuan University from January 2020 to December 2023

Exclusion Criteria:

* Under the age of 18;
* Gender unknown;
* Incorrect or invalid discharge diagnosis;
* The hospitalization time is less than 24 hours;
* Data information is missing by more than 30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of clinical data of patients diagnosed with sepsis at West China Hospital of Sichuan University from January 2020 to December 2023. Review and summarize the baseline data of patients (including age, gender, comorbidities, history of malignant tumors, lesion location, pathological type, etc.), occurrence of serious complications, total length of hospital stay, survival time, and construct a time-series based mortality risk prognosis prediction model for sepsis patients.
Sampling Method: Non-Probability Sample
Enrollment: 3641 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Biomarker level | 5 Years
  Including inflammatory markers (such as C-reactive protein (CRP), interleukins (IL-6, IL-10), and procalcitonin (PCT)) and metabolic markers (such as lactate levels and arterial blood gas pH values) for sepsis prognostic analysis.

SECONDARY OUTCOMES:
SOFA score | 5 Years
  Standard measure of organ function for sepsis.
Length of ICU stay | 5 Years
  Reflects the severity of illness and critical care needs.
APACHE II score | 5 Years
  Standard measure of severity for sepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Zhang, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided